CLINICAL TRIAL: NCT06162286
Title: A Phase 3b Randomized, Double-blind, Multi-center Study to Compare the Safety and Efficacy of Omadacycline IV/PO to Moxifloxacin IV/PO for Treating Adult Subjects With Community-acquired Bacterial Pneumonia (CABP)
Brief Title: A Phase 3b Randomized, Double-blind, Multi-center Study to Compare the Safety and Efficacy of Omadacycline to Moxifloxacin for Treating Adult Subjects With CABP
Acronym: public
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zai Lab (Hong Kong), Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZL-2401-004
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Community-acquired Bacterial Pneumonia
MeSH Terms: interventions — omadacycline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxifloxacin (Active Comparator): Moxifloxacin IV/PO
  Interventions: Drug: Moxifloxacin
- Omadacycline (Experimental): Omadacycline IV/PO
  Interventions: Drug: Omadacycline

INTERVENTIONS:
Drug: Omadacycline — Omadacycline IV/PO
  Arms: Omadacycline
Drug: Moxifloxacin — Moxifloxacin IV/PO
  Arms: Moxifloxacin

SUMMARY:
The primary objective of the study is to show that in Chinese adults with CABP, a course of IV/PO treatment with omadacycline has similar clinical efficacy as the with the comparator antibiotic, IV/PO moxifloxacin. The study is designed as a bridging study, to confirm the results of the pivotal global CABP trial in an ethnically different population of Chinese.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent obtained before any protocol specific assessment is performed.
2. Male or female, ages 18 years or older.
3. Has at least 3 of the following symptoms:

   * Cough
   * Production of purulent sputum
   * Dyspnea (shortness of breath)
   * Chest pain
4. Has at least 2 of the following abnormal vital signs:

   * Fever or hypothermia documented by the investigator (temperature > 38.0°C or < 36.0°C)
   * Hypotension with systolic blood pressure (SBP) < 90 mmHg
   * Heart rate (HR) > 90 beats per minute (bpm)
   * Respiratory rate (RR) > 20 breaths/minute

Exclusion Criteria:

1. Has received antibacterial treatment >24hr within the 72hr window prior to randomization.

   Subjects may be eligible despite prior antibacterial therapy if they had been treated with short action time antimicrobial for ≤24h, or if they have received > 48 hours of prior systemic antibacterial therapy for the current episode of CABP with unequivocal clinical evidence of treatment failure.
2. Is known or suspected to have CABP caused by a pathogen that may be resistant to either test article (eg, Klebsiella pneumoniae, Pseudomonas aeruginosa, Pneumocystis jiroveci, obligate anaerobes, mycobacteria, fungal pathogens).
3. Suspected or confirmed empyema (a parapneumonic pleural effusion is not an exclusion criteria) or lung abscess.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall assessment of clinical response rate at post therapy evaluation (PTE) timepoint in the mITT population. | 18 months

SECONDARY OUTCOMES:
Clinical response rate at the Early Clinical Response (ECR) assessment (72 to 120 hours after administration of the first dose of test article) in the mITT population. | 72 to 120 hours
Clinical response rate at the End of Treatment (EOT) assessment in the mITT and CE population. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Haihui Huang, PhD, Principal Investigator — Huashan Hospital
Locations (40):
- China (40):
  - Beijing Tsinghua Chang Gung Hospital/Infectious Diseases Department, Beijing
  - Peking University Shougang Hospital/Respiratory and Critical Care Medicine Department, Beijing
  - The First Affiliated Hospital of Bengbu Medical College/Intensive care unit, Bengbu
  - The Central Hospital of Changsha/Department of Respiratory and Critical Care Medicine, Changsha
  - The Third Hospital of Changsha/Respiratory and Critical Care Medicine Department, Changsha
  - Xiangya Hospital Central South University/Department of Respiratory and Critical Care Medicine, Changsha
  - West China Hospital of Sichuan University/Infectious Disease Center, Chengdu
  - The First People's Hospital of Foshan/Department of Respiratory and Critical Care Medicine, Foshan
  - Fuyang People's Hospital/Department of Respiratory and Critical Care Medicine, Fuyang
  - The First Affiliated Hospital of Gannan Medical University/Pneumology Department, Gannan
  - Guangdong Second Central Hospital/Department of Respiratory and Critical Care Medicine, Guangzhou
  - Guangzhou First People's Hospital/Respiratory and Critical Care Medicine Department, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University/Respiratory Medicine, Guangzhou
  - The Hospital of Zhejiang/Respiratory Medicine, Hangzhou
  - Jiangyin People's Hospital/Department of Respiratory and Critical Care Medicine, Jiangyin
  - The First Hospital of Jiaxing/Pneumology Department, Jiaxing
  - Kunming First People's Hospital/Respiratory Medicine, Kunming
  - The Central Hospital of Luoyang/Department of Respiratory and Critical Care Medicine, Luoyang
  - The Central Hospital of Mianyang/Department of Respiratory and Critical Care Medicine, Mianyang
  - Jiangxi Province People's Hospital/Pneumology Department, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First People's Hospital of Nanning/Department of Respiratory and Critical Care Medicine, Nanning
  - The People's Hospital of Guangxi Zhuang Autonomous Region/Department of Respiratory and Critical Care Medicine, Nanning
  - Quanzhou First Hospital/Infectious Disease Department, Quanzhou
  - Huashan Hospital, Shanghai
  - Shanghai Fifth People's Hospital,Fudan University/Department of Respiratory and Critical Care Medicine, Shanghai
  - Shanghai Pulmonary Hospital/Respiratory and Critical Care Medicine Department, Shanghai
  - The Central Hospital of Shenyang/Department of Respiratory and Critical Care Medicine, Shenyang
  - Shenzhen People's Hospital/Department of Respiratory and Critical Care Medicine, Shenzhen
  - Shijiazhuang People's Hospital/Respiratory Medicine, Shijia Zhuang
  - Suzhou Municipal Hospital/Department of Respiratory and Critical Care Medicine, Suzhou
  - The 2nd Affiliated Hospital of Wenzhou Medical University/Department of Respiratory and Critical Care Medicine, Wenzhou
  - Wenzhou Central Hospital/Department of Respiratory and Critical Care Medicine, Wenzhou
  - The Central Hospital of Wuhan/Respiratory and Critical Care Medicine Department, Wuhan
  - Zhongshan Hospital Xiamen University/Pneumology Department, Xiamen
  - The First Affiliated Hospital of Xinjiang Medical University/Pneumology Department, Xinjiang
  - The Central Hospital of Xinxiang/Department of Respiratory and Critical Care Medicine, Xinxiang
  - People's Hospital of Ningxia Hui Autonomous Region/Pneumology Department, Yinchuan
  - Zhejiang Provincial People's Hospital/Respiratory Medicine, Zhejiang
  - Zibo Municipal Hospital/Department of Respiratory and Critical Care Medicine, Zibo